CLINICAL TRIAL: NCT00714077
Title: Prospective Randomized Phase III Study of Concurrent Capecitabine and Radiotherapy With or Without Oxaliplatin as Adjuvant Treatment for Stage II and III Rectal Cancer
Brief Title: Adjuvant Treatment of Concurrent RT and CAPOX or Capecitabine Alone for Stage II and III Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Cancer Hospital of Guizhou Province (Other); Shandong Cancer Hospital and Institute (Other); Hebei Medical University Fourth Hospital (Other); Peking University Third Hospital (Other); General Hospital of Chinese Armed Police Forces (Other); Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Jing Jin, M.D., M.D., Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: CAMS_rectal cancer_01
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Rectal Neoplasms
Keywords: rectal cancer; concurrent chemoradiotherapy; adjuvant therapy; phase III study
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- adjuvant capecitabine: To compare different adjuvant concurrent chemoradiotherapy regimen (Oxaliplatin with capecitabine vs capecitabine) for patients with II/III rectal cancer
- adjuvant oxaliplatin and capecitabine: To compare different adjuvant concurrent chemoradiotherapy regimen (Oxaliplatin with capecitabine vs capecitabine) for patients with II/III rectal cancer

SUMMARY:
The purpose of this study is:

* To compare the long-term of survival and local/regional control between the two postoperative concurrent chemoradiotherapy regimens: capecitabine vs. oxaliplatin and capecitabine,for stage II and III rectal cancer
* To compare the toxicity profile between the two different concurrent chemoradiotherapy regimens.

DETAILED DESCRIPTION:
Adjuvant 5-FU based concurrent chemoradiotherapy and chemotherapy is the standard care for locally advanced stage II-III rectal cancer, based on several randomized Phase III clinical trials. With this standard treatment, 5-year local failure rate and distant metastasis rate is 10% and around 35%, respectively. Capecitabine, an analog of 5-fluoruracil (5FU), was demonstrated to have similar treatment results compared to 5-FU, but have much lower toxicities. Oxaliplatin based chemotherapy, also showed a better disease-free survival rate compared with 5-FU based-regimen. So far, some Phase I/II studies have shown the safety and preliminary results of either concurrent chemotherapy of capecitabine or oxaliplatin and capecitabine. The long-term results in comparison of capecitabine concurrent chemoradiotherapy with oxaliplatin/capecitabine concurrent chemoradiotherapy need to be further analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old,male or female
* R0 surgery
* Pathologically approved as stage II or stage III
* Enrolled within 6 months from the date of surgery
* Upper border of tumor before surgery was under L5
* KPS>70% or ECOG 0-2
* No prior radiotherapy in the past 6 months
* Received chemotherapy no more than 4 cycles after surgery
* HGB>100 g/L, WBC≥3.5x109 /L, PLT≥100x109 /L; CR<1.5 x Upper normality，TB<2.5 X Upper normality，AST or ALT<2.5 x Upper normality，AKP<2.5 X Upper normality
* Signed consent

Exclusion Criteria:

* Other malignancies simultaneously except in situ cervix or nonmelanoma skin cancer
* Pregnancy or in lactation
* HGB<100 g/L, WBC<3.5x109 /L, PLT<100x109 /L; CR≥1.5 x Upper normality，TB≥2.5 X Upper normality，AST or ALT≥2.5 x Upper normality，AKP≥2.5 X Upper normality

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicenter patients enrollment
Sampling Method: Probability Sample
Enrollment: 570 (Estimated)
Dates: Start 2008-04; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | the day of surgery to the date of the event

SECONDARY OUTCOMES:
overall survival rate | the day of surgery to the date of death or last follow-up
cumulative incidence of local recurrence | the day of surgery to the date of local recurrence
cumulative incidence of distant metastasis | the day of surgery to the date of distant metastasis
compliance | during adjuvant radiotherapy and chemotherapy
safety | the day of randomization to the date of death or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yexiong Li, M.D., Principal Investigator — CAMS; Jing Jin, M.D.;Ph.D, Principal Investigator — CAMS
Locations (1):
- Jing Jin, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Tveit KM, Guldvog I, Hagen S, Trondsen E, Harbitz T, Nygaard K, Nilsen JB, Wist E, Hannisdal E. Randomized controlled trial of postoperative radiotherapy and short-term time-scheduled 5-fluorouracil against surgery alone in the treatment of Dukes B and C rectal cancer. Norwegian Adjuvant Rectal Cancer Project Group. Br J Surg. 1997 Aug;84(8):1130-5. PMID 9278661
- [Background] Wolmark N, Wieand HS, Hyams DM, Colangelo L, Dimitrov NV, Romond EH, Wexler M, Prager D, Cruz AB Jr, Gordon PH, Petrelli NJ, Deutsch M, Mamounas E, Wickerham DL, Fisher ER, Rockette H, Fisher B. Randomized trial of postoperative adjuvant chemotherapy with or without radiotherapy for carcinoma of the rectum: National Surgical Adjuvant Breast and Bowel Project Protocol R-02. J Natl Cancer Inst. 2000 Mar 1;92(5):388-96. doi: 10.1093/jnci/92.5.388. PMID 10699069
- [Background] Gastrointestinal Tumor Study Group. Prolongation of the disease-free interval in surgically treated rectal carcinoma. N Engl J Med. 1985 Jun 6;312(23):1465-72. doi: 10.1056/NEJM198506063122301. PMID 2859523
- [Background] Krook JE, Moertel CG, Gunderson LL, Wieand HS, Collins RT, Beart RW, Kubista TP, Poon MA, Meyers WC, Mailliard JA, et al. Effective surgical adjuvant therapy for high-risk rectal carcinoma. N Engl J Med. 1991 Mar 14;324(11):709-15. doi: 10.1056/NEJM199103143241101. PMID 1997835
- [Background] de Gramont A, Figer A, Seymour M, Homerin M, Hmissi A, Cassidy J, Boni C, Cortes-Funes H, Cervantes A, Freyer G, Papamichael D, Le Bail N, Louvet C, Hendler D, de Braud F, Wilson C, Morvan F, Bonetti A. Leucovorin and fluorouracil with or without oxaliplatin as first-line treatment in advanced colorectal cancer. J Clin Oncol. 2000 Aug;18(16):2938-47. doi: 10.1200/JCO.2000.18.16.2938. PMID 10944126
- [Background] Giacchetti S, Perpoint B, Zidani R, Le Bail N, Faggiuolo R, Focan C, Chollet P, Llory JF, Letourneau Y, Coudert B, Bertheaut-Cvitkovic F, Larregain-Fournier D, Le Rol A, Walter S, Adam R, Misset JL, Levi F. Phase III multicenter randomized trial of oxaliplatin added to chronomodulated fluorouracil-leucovorin as first-line treatment of metastatic colorectal cancer. J Clin Oncol. 2000 Jan;18(1):136-47. doi: 10.1200/JCO.2000.18.1.136. PMID 10623704
- [Background] Andre T, Boni C, Mounedji-Boudiaf L, Navarro M, Tabernero J, Hickish T, Topham C, Zaninelli M, Clingan P, Bridgewater J, Tabah-Fisch I, de Gramont A; Multicenter International Study of Oxaliplatin/5-Fluorouracil/Leucovorin in the Adjuvant Treatment of Colon Cancer (MOSAIC) Investigators. Oxaliplatin, fluorouracil, and leucovorin as adjuvant treatment for colon cancer. N Engl J Med. 2004 Jun 3;350(23):2343-51. doi: 10.1056/NEJMoa032709. PMID 15175436
- [Background] Van Cutsem E, Hoff PM, Harper P, Bukowski RM, Cunningham D, Dufour P, Graeven U, Lokich J, Madajewicz S, Maroun JA, Marshall JL, Mitchell EP, Perez-Manga G, Rougier P, Schmiegel W, Schoelmerich J, Sobrero A, Schilsky RL. Oral capecitabine vs intravenous 5-fluorouracil and leucovorin: integrated efficacy data and novel analyses from two large, randomised, phase III trials. Br J Cancer. 2004 Mar 22;90(6):1190-7. doi: 10.1038/sj.bjc.6601676. PMID 15026800
- [Background] Twelves C, Wong A, Nowacki MP, Abt M, Burris H 3rd, Carrato A, Cassidy J, Cervantes A, Fagerberg J, Georgoulias V, Husseini F, Jodrell D, Koralewski P, Kroning H, Maroun J, Marschner N, McKendrick J, Pawlicki M, Rosso R, Schuller J, Seitz JF, Stabuc B, Tujakowski J, Van Hazel G, Zaluski J, Scheithauer W. Capecitabine as adjuvant treatment for stage III colon cancer. N Engl J Med. 2005 Jun 30;352(26):2696-704. doi: 10.1056/NEJMoa043116. PMID 15987918
- [Background] Sawada N, Ishikawa T, Sekiguchi F, Tanaka Y, Ishitsuka H. X-ray irradiation induces thymidine phosphorylase and enhances the efficacy of capecitabine (Xeloda) in human cancer xenografts. Clin Cancer Res. 1999 Oct;5(10):2948-53. PMID 10537364
- [Background] Cividalli A, Ceciarelli F, Livdi E, Altavista P, Cruciani G, Marchetti P, Danesi DT. Radiosensitization by oxaliplatin in a mouse adenocarcinoma: influence of treatment schedule. Int J Radiat Oncol Biol Phys. 2002 Mar 15;52(4):1092-8. doi: 10.1016/s0360-3016(01)02792-4. PMID 11958906
- [Background] Kim JC, Kim TW, Kim JH, Yu CS, Kim HC, Chang HM, Ryu MH, Park JH, Ahn SD, Lee SW, Shin SS, Kim JS, Choi EK. Preoperative concurrent radiotherapy with capecitabine before total mesorectal excision in locally advanced rectal cancer. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):346-53. doi: 10.1016/j.ijrobp.2005.02.046. PMID 15913913
- [Background] Kuebler JP, Wieand HS, O'Connell MJ, Smith RE, Colangelo LH, Yothers G, Petrelli NJ, Findlay MP, Seay TE, Atkins JN, Zapas JL, Goodwin JW, Fehrenbacher L, Ramanathan RK, Conley BA, Flynn PJ, Soori G, Colman LK, Levine EA, Lanier KS, Wolmark N. Oxaliplatin combined with weekly bolus fluorouracil and leucovorin as surgical adjuvant chemotherapy for stage II and III colon cancer: results from NSABP C-07. J Clin Oncol. 2007 Jun 1;25(16):2198-204. doi: 10.1200/JCO.2006.08.2974. Epub 2007 Apr 30. PMID 17470851
- [Background] Jin J, Li YX, Liu YP, Wang WH, Song YW, Li T, Li N, Yu ZH, Liu XF. A phase I study of concurrent radiotherapy and capecitabine as adjuvant treatment for operable rectal cancer. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):725-9. doi: 10.1016/j.ijrobp.2005.08.017. Epub 2005 Oct 19. PMID 16242260
- [Background] Souglakos J, Androulakis N, Mavroudis D, Kourousis C, Kakolyris S, Vardakis N, Kalbakis K, Pallis A, Ardavanis A, Varveris C, Georgoulias V. Multicenter dose-finding study of concurrent capecitabine and radiotherapy as adjuvant treatment for operable rectal cancer. Int J Radiat Oncol Biol Phys. 2003 Aug 1;56(5):1284-7. doi: 10.1016/s0360-3016(03)00275-x. PMID 12873672
- [Background] Ngan SY, Michael M, Mackay J, McKendrick J, Leong T, Lim Joon D, Zalcberg JR. A phase I trial of preoperative radiotherapy and capecitabine for locally advanced, potentially resectable rectal cancer. Br J Cancer. 2004 Sep 13;91(6):1019-24. doi: 10.1038/sj.bjc.6602106. PMID 15305186
- [Background] Dunst J, Reese T, Sutter T, Zuhlke H, Hinke A, Kolling-Schlebusch K, Frings S. Phase I trial evaluating the concurrent combination of radiotherapy and capecitabine in rectal cancer. J Clin Oncol. 2002 Oct 1;20(19):3983-91. doi: 10.1200/JCO.2002.02.049. PMID 12351595
- [Background] Rodel C, Grabenbauer GG, Papadopoulos T, Hohenberger W, Schmoll HJ, Sauer R. Phase I/II trial of capecitabine, oxaliplatin, and radiation for rectal cancer. J Clin Oncol. 2003 Aug 15;21(16):3098-104. doi: 10.1200/JCO.2003.02.505. PMID 12915600
- [Background] Fakih MG, Rajput A, Yang GY, Pendyala L, Toth K, Smith JL, Lawrence DD, Rustum YM. A Phase I study of weekly intravenous oxaliplatin in combination with oral daily capecitabine and radiation therapy in the neoadjuvant treatment of rectal adenocarcinoma. Int J Radiat Oncol Biol Phys. 2006 Aug 1;65(5):1462-70. doi: 10.1016/j.ijrobp.2006.03.003. Epub 2006 Jun 5. PMID 16750332
- [Background] Glynne-Jones R, Sebag-Montefiore D, Maughan TS, Falk SJ, McDonald AC. A phase I dose escalation study of continuous oral capecitabine in combination with oxaliplatin and pelvic radiation (XELOX-RT) in patients with locally advanced rectal cancer. Ann Oncol. 2006 Jan;17(1):50-6. doi: 10.1093/annonc/mdj031. Epub 2005 Nov 10. PMID 16284060
- [Background] Machiels JP, Duck L, Honhon B, Coster B, Coche JC, Scalliet P, Humblet Y, Aydin S, Kerger J, Remouchamps V, Canon JL, Van Maele P, Gilbeau L, Laurent S, Kirkove C, Octave-Prignot M, Baurain JF, Kartheuser A, Sempoux C. Phase II study of preoperative oxaliplatin, capecitabine and external beam radiotherapy in patients with rectal cancer: the RadiOxCape study. Ann Oncol. 2005 Dec;16(12):1898-905. doi: 10.1093/annonc/mdi406. Epub 2005 Oct 11. PMID 16219623
- [Background] Schmoll HJ, Cartwright T, Tabernero J, Nowacki MP, Figer A, Maroun J, Price T, Lim R, Van Cutsem E, Park YS, McKendrick J, Topham C, Soler-Gonzalez G, de Braud F, Hill M, Sirzen F, Haller DG. Phase III trial of capecitabine plus oxaliplatin as adjuvant therapy for stage III colon cancer: a planned safety analysis in 1,864 patients. J Clin Oncol. 2007 Jan 1;25(1):102-9. doi: 10.1200/JCO.2006.08.1075. PMID 17194911
- [Background] De Paoli A, Chiara S, Luppi G, Friso ML, Beretta GD, Del Prete S, Pasetto L, Santantonio M, Sarti E, Mantello G, Innocente R, Frustaci S, Corvo R, Rosso R. Capecitabine in combination with preoperative radiation therapy in locally advanced, resectable, rectal cancer: a multicentric phase II study. Ann Oncol. 2006 Feb;17(2):246-51. doi: 10.1093/annonc/mdj041. Epub 2005 Nov 9. PMID 16282246
- [Background] Rodel F, Hoffmann J, Grabenbauer GG, Papadopoulos T, Weiss C, Gunther K, Schick C, Sauer R, Rodel C. High survivin expression is associated with reduced apoptosis in rectal cancer and may predict disease-free survival after preoperative radiochemotherapy and surgical resection. Strahlenther Onkol. 2002 Aug;178(8):426-35. doi: 10.1007/s00066-002-1003-y. PMID 12240548
- [Background] Ruzzo A, Graziano F, Loupakis F, Rulli E, Canestrari E, Santini D, Catalano V, Ficarelli R, Maltese P, Bisonni R, Masi G, Schiavon G, Giordani P, Giustini L, Falcone A, Tonini G, Silva R, Mattioli R, Floriani I, Magnani M. Pharmacogenetic profiling in patients with advanced colorectal cancer treated with first-line FOLFOX-4 chemotherapy. J Clin Oncol. 2007 Apr 1;25(10):1247-54. doi: 10.1200/JCO.2006.08.1844. PMID 17401013
- [Background] Gordon MA, Gil J, Lu B, Zhang W, Yang D, Yun J, Schneider S, Groshen S, Iqbal S, Press OA, Rhodes K, Lenz HJ. Genomic profiling associated with recurrence in patients with rectal cancer treated with chemoradiation. Pharmacogenomics. 2006 Jan;7(1):67-88. doi: 10.2217/14622416.7.1.67. PMID 16354126
- [Background] Stoehlmacher J, Park DJ, Zhang W, Yang D, Groshen S, Zahedy S, Lenz HJ. A multivariate analysis of genomic polymorphisms: prediction of clinical outcome to 5-FU/oxaliplatin combination chemotherapy in refractory colorectal cancer. Br J Cancer. 2004 Jul 19;91(2):344-54. doi: 10.1038/sj.bjc.6601975. PMID 15213713
- [Derived] Li N, Zhu Y, Liu LY, Feng YR, Wang WL, Wang J, Wang H, Li GF, Tang Y, Hu C, Liu WY, Ren H, Wang SL, Wang WH, Song YW, Liu YP, Fang H, Tang Y, Lu NN, Chen B, Qi SN, Liu XF, Li YX, Jin J. Postoperative Chemoradiotherapy With Capecitabine and Oxaliplatin vs Capecitabine for Stage II to III Rectal Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2021 Nov 1;4(11):e2136116. doi: 10.1001/jamanetworkopen.2021.36116. PMID 34846525